CLINICAL TRIAL: NCT03013257
Title: A Randomized, Open-label, Parallel-group Study to Explore the Efficacy of High-intensity Focused Ultrasound (HIFU) Versus Fixed-dose Radioiodine-131 in the Treatment of Relapsed Graves' Disease
Brief Title: HIFU vs RAI in the Relapsed Graves' Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Lang Hung Hin, Brian, Clinical Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UW 16-565
Record Dates: First submitted 2017-01-04; First posted 2017-01-06 (Estimated); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Graves Disease
Keywords: Relapsed Graves' disease; High Intensity Focused Ultrasound; RAI
MeSH Terms: conditions — Graves Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Intensity Focused Ultrasound (Experimental): Try to use the machine 'Echopulse' with High Intensity Focused Ultrasound to treat the relapsed Graves' disease
  Interventions: Device: Echopulse
- Fixed-dose radioiodine-131 (No Intervention): Using the traditional treatment, fixed-dose radioiodine-131, to treat the relapsed Graves' disease

INTERVENTIONS:
Device: Echopulse — Replacing HIFU for the Graves' disease patients who traditionally have RAI to remission
  Other Names: High Intensity Focused Ultrasound (HIFU)
  Arms: High Intensity Focused Ultrasound

SUMMARY:
Graves' disease (GD) is an autoimmune thyroid disorder caused by stimulating auto-antibodies to the thyrotrophin (TSH) receptor on thyroid follicular cells. It is the most common cause of hyperthyroidism and approximately 3% of women and 0.5% of men develop GD in their lifetime.

RAI has been shown to be a cost-effective and safe therapy in patients with GD but with some disadvantages. In addition, despite its proven efficacy and safety, many patients do not wish to undergo RAI because of radiation fear and prefer to either continue ATDs or have surgery.

High-intensity focused ultrasound (HIFU) is a non-invasive procedure that involves the application of a high-energy focused beam for thermal tissue ablation within a targeted zone. Similar to the principle of RAI (i.e. using ionizing radiation to ablate thyroid parenchyma and cause GD remission), we postulated that the heat energy generated from HIFU could also be used to ablate the thyroid parenchyma and cause GD remission. The idea of using heat energy to ablate thyroid parenchyma minimally invasively was recently reported using radiofrequency ablation but to our knowledge, we are one of the first (if not the first) group to propose using HIFU energy to ablate thyroid parenchyma as a definitive treatment for relapsed GD.

Having obtained ethical approval, a pilot study was conducted to examine the efficacy and safety of HIFU as a treatment for relapsed GD. In the pilot study, all patients underwent a safe and successful HIFU ablation for relapsed GD. Based on the results of the pilot study, we hypothesize that a single HIFU treatment to the thyroid gland may be as effective as our standard outpatient fixed-dose of RAI (370MBq) in causing remission of GD at 6-month. If our hypothesis turns out to be true, HIFU could become a treatment option for patients who are indicated for RAI but do not wish to have it because of one reason or another. HIFU appears to induce a faster disease remission and lessen the need of deferring pregnancy and radiation precautions because of the absence of radioactivity.

DETAILED DESCRIPTION:
Graves' disease (GD) is an autoimmune thyroid disorder caused by stimulating auto-antibodies to the thyrotrophin (thyroid stimulating hormone [TSH]) receptor on thyroid follicular cells. It is the most common cause of hyperthyroidism and approximately 3% of women and 0.5% of men develop GD in their lifetime1. In our locality, like Europe and Japan, antithyroid drugs (ATDs) such as carbimazole or propylthiouracil have been preferred over radioactive iodine (RAI) and surgery as the initial treatment of GD2-4. This is because ATDs are relatively easy to administer, could induce disease remission (30-70%) and avoid life-long thyroid hormone replacement, operative risks and radioactivity2-4. However, because of possible side-effects, they are only recommended for a period of 12 to 18 months. Taking ATDs for a longer period does not seem to increase the chance of remission5. Therefore, currently, once the disease has relapsed after a 18-month of ATD treatment, more definitive treatment modalities like RAI or surgery are indicated. Regarding to which is more preferable, surgery is usually advised in patients with large compressive goiter (>80g), suspected or documented thyroid malignancy, planning to become pregnant within 6 months and moderate to severe Graves' ophthalmopathy (GO)2-4. As a result, most patients without these conditions are considered for RAI2-4.

RAI has been shown to be a cost-effective and safe therapy in patients with GD4,6,7. In North America, clinical endocrinologists favor RAI as the initial treatment for GD2-4. However, since RAI is usually prescribed on an outpatient basis, it is necessary to consider nearby individuals' exposure doses and formulate radiation precautions carefully8. Other disadvantages include its slow induction of euthyroidism, potential worsening of GO and deferral of pregnancy2-4. Although various dosing techniques have been described to ensure an adequate radiation delivery to the thyroid gland, the simplest and most effective method has been to administer a fixed dose of RAI2. However, due to local regulations and our densely-populated areas, administering higher RAI doses (>400MBq) is not permitted on an outpatient basis9. As a result, the usual RAI dose usually ranges between 185 to 370MBq (i.e. up to 10mci)10. In addition, despite its proven efficacy and safety, many patients do not wish to undergo RAI because of radiation fear and prefer to either continue ATDs or have surgery11.

High-intensity focused ultrasound (HIFU) is a non-invasive procedure that involves the application of a high-energy focused beam for thermal tissue ablation within a targeted zone. It has been applied in a variety of medical conditions including uterine fibroids and prostate, breast, pancreatic, and liver tumors12. Unlike other ablation devices (like radiofrequency or laser ablation), HIFU does not require needle puncture and is considered safer and less operator-dependent13. Single HIFU treatment has been shown to reduce size of benign thyroid nodules13,14. Histologic examination confirmed that HIFU induced complete tissue necrosis within a targeted area13. Similar to the principle of RAI (i.e. using ionizing radiation to ablate thyroid parenchyma and cause GD remission), we postulated that the heat energy generated from HIFU could also be used to ablate the thyroid parenchyma and cause GD remission. The idea of using heat energy to ablate thyroid parenchyma minimally invasively was recently reported using radiofrequency ablation15 but to our knowledge, we are one of the first (if not the first) group to propose using HIFU energy to ablate thyroid parenchyma as a definitive treatment for relapsed GD.

Having obtained ethical approval, a pilot study was conducted to examine the efficacy and safety of HIFU as a treatment for relapsed GD. Over a 2-month period, 20 patients underwent a single HIFU treatment for relapsed GD. The treatment involved ablating the entire right, left and central (isthmic) lobes with HIFU pulses. To avoid inadvertent injury to heat-sensitive structures like the recurrent laryngeal nerve, parathyroid glands, trachea and esophagus, we deliberately left 2-3ml of thyroid parenchyma non-ablated close to the trachea-esophageal groove on each side. The reason for not leaving a larger amount of non-ablated parenchyma is because from the experience in subtotal thyroidectomy, leaving > 6ml of normal parenchyma may diminish the long-term remission rate16.

In the pilot study, all patients underwent a safe and successful HIFU ablation for relapsed GD. By ultrasound (USG) volumetry, the mean pre-ablation total thyroid volume was 18.5 ± 6.4ml. The average treatment time was 72.7 ± 31.0 mins and the total energy delivered to each patient was 21.4 ± 5.9 KJ. No patients suffered any major complications afterwards except for 2 patients (10.0%) who had minor neck redness in the first week. By 4-week, all patients were either biochemically euthyroid (n=15) (without ATDs) or biochemically hypothyroid (requiring thyroxine replacement) (n=5). At 6-month, 15 (75.0%) patients remained biochemically euthyroid or hypothyroid without ATDs (i.e. remission) while 5 patients (25.0%) had biochemical hyperthyroidism. However, of these, only 3 required ATDs and 2 were kept observed.

Based on the results of the pilot study, we hypothesize that a single HIFU treatment to the thyroid gland may be as effective as our standard outpatient fixed-dose of RAI (370MBq) in causing remission of GD at 6-month. If our hypothesis turns out to be true, HIFU could become a treatment option for patients who are indicated for RAI but do not wish to have it because of one reason or another. Apart from the benefit of being an outpatient treatment, HIFU appears to induce a faster disease remission and lessen the need of deferring pregnancy and radiation precautions because of the absence of radioactivity.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of GD based on standard clinical criteria (elevated thyroid hormone levels, suppressed TSH, positive TSHR auto-antibody, diffuse goiter ± high RAI uptake).
2. Aged between 18 and 70 years old at the time of informed consent
3. Have had at least one GD relapse. A relapse is defined as recurrent or persistent hyperthyroidism despite completing a continued course of ATDs for 18 months or more.
4. Indicated for RAI treatment
5. Valid consent is obtained

Exclusion Criteria:

1. Prefer or have clear indications for surgery (such as those with large compressive goiter, suspected or documented thyroid malignancy, wishing to become pregnant within 6 months or with moderate to severe GO).
2. Have pre-existing vocal cord palsy
3. Are unable to move or extend their neck
4. Have either right, left or central (isthmic) lobe measuring >30ml in volume on pre-treatment USG volumetry (see later)
5. Have concomitant thyroid nodules which are either indeterminate, suspicious of malignancy or proven malignant on fine needle aspiration cytology (FNAC).
6. Have active or severe Graves ophthalmopathy (GO)
7. Are pregnant, lactating or planning for pregnancy within 6 months
8. Have any medical conditions that would make them too ill to undergo intravenous sedation or treatment
9. Any condition that is unstable or can jeopardize the safety of the patients and their compliance to the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2017-04-25 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Rate of remission | 6 months
  Stating of biochemically euthyroid and hypothyroid without ATDs after 6 months of treatment

SECONDARY OUTCOMES:
Incidence of treatment-related morbidities from day-0 to post 2-week | 2 weeks
  To examine any treatment-related morbidities after the treatment within 2 weeks.
Change in auto-antibodies | 6 months
  To examine the changes of anti-thyroid and TSHR after 6 months of treatment
Change in total thyroid volume | 6 months
  To measure the change in size of total thyroid volume after 6 months of treatment
Change in eye disease activity | 6 months
  To examine the change in eye disease activity (CAS) with 6 months.
Satisfaction score after treatment | 6 months
  To measure the satisfaction score (1-10) after treatment
The pain assessment after treatment | 6 months
  The pain assessment (scoring 1-10) after treatment
Change in Quality of life | 6 months
  To examine the change in qualitfy of life with SF-12 scores from baseline to 2-month and 6-month
The medical costs | 6 months
  To evaluate the cost of different treatments including direct medical costs (including treatment, investigations, unplanned readmission and visits) and indirect costs (such as number of days before returning to normal activities and work). Medical costs will be based on the latest Government Gazette.
The effectiveness of HIFU treatment | 6 months
  The effectiveness of HIFU will be quantified by quality-adjusted left years (QALYs), which will be calculated as the product of the average duration of that stage and SF-6D preference value (i.e. from SF-12) for the particular health state.

CONTACTS AND LOCATIONS:
Overall Officials: Hung Hin, Brian Lang, MBBS(Hons), Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nystrom HF, Jansson S, Berg G. Incidence rate and clinical features of hyperthyroidism in a long-term iodine sufficient area of Sweden (Gothenburg) 2003-2005. Clin Endocrinol (Oxf). 2013 May;78(5):768-76. doi: 10.1111/cen.12060. PMID 23421407
- [Background] Bahn Chair RS, Burch HB, Cooper DS, Garber JR, Greenlee MC, Klein I, Laurberg P, McDougall IR, Montori VM, Rivkees SA, Ross DS, Sosa JA, Stan MN; American Thyroid Association; American Association of Clinical Endocrinologists. Hyperthyroidism and other causes of thyrotoxicosis: management guidelines of the American Thyroid Association and American Association of Clinical Endocrinologists. Thyroid. 2011 Jun;21(6):593-646. doi: 10.1089/thy.2010.0417. Epub 2011 Apr 21. PMID 21510801
- [Background] Burch HB, Cooper DS. Management of Graves Disease: A Review. JAMA. 2015 Dec 15;314(23):2544-54. doi: 10.1001/jama.2015.16535. PMID 26670972
- [Background] Franklyn JA, Boelaert K. Thyrotoxicosis. Lancet. 2012 Mar 24;379(9821):1155-66. doi: 10.1016/S0140-6736(11)60782-4. Epub 2012 Mar 5. PMID 22394559
- [Background] Abraham P, Avenell A, Park CM, Watson WA, Bevan JS. A systematic review of drug therapy for Graves' hyperthyroidism. Eur J Endocrinol. 2005 Oct;153(4):489-98. doi: 10.1530/eje.1.01993. PMID 16189168
- [Background] Sundaresh V, Brito JP, Wang Z, Prokop LJ, Stan MN, Murad MH, Bahn RS. Comparative effectiveness of therapies for Graves' hyperthyroidism: a systematic review and network meta-analysis. J Clin Endocrinol Metab. 2013 Sep;98(9):3671-7. doi: 10.1210/jc.2013-1954. Epub 2013 Jul 3. PMID 23824415
- [Background] Patel NN, Abraham P, Buscombe J, Vanderpump MP. The cost effectiveness of treatment modalities for thyrotoxicosis in a U.K. center. Thyroid. 2006 Jun;16(6):593-8. doi: 10.1089/thy.2006.16.593. PMID 16839261
- [Background] Liu B, Tian R, Peng W, He Y, Huang R, Kuang A. Radiation Safety Precautions in (131)I Therapy of Graves' Disease Based on Actual Biokinetic Measurements. J Clin Endocrinol Metab. 2015 Aug;100(8):2934-41. doi: 10.1210/jc.2015-1682. Epub 2015 Jun 5. PMID 26046966
- [Background] Yau JS, Chu KS, Li JK, Chan KW, Lau IT, Yum SW, Chan CW, Mo LK, Kwan WK. Usage of a fixed dose of radioactive iodine for the treatment of hyperthyroidism: one-year outcome in a regional hospital in Hong Kong. Hong Kong Med J. 2009 Aug;15(4):267-73. PMID 19652233
- [Background] Yip J, Lang BH, Lo CY. Changing trend in surgical indication and management for Graves' disease. Am J Surg. 2012 Feb;203(2):162-7. doi: 10.1016/j.amjsurg.2011.01.029. Epub 2011 Jun 17. PMID 21683939
- [Background] Zhou YF. High intensity focused ultrasound in clinical tumor ablation. World J Clin Oncol. 2011 Jan 10;2(1):8-27. doi: 10.5306/wjco.v2.i1.8. PMID 21603311
- [Background] Esnault O, Franc B, Chapelon JY. Localized ablation of thyroid tissue by high-intensity focused ultrasound: improvement of noninvasive tissue necrosis methods. Thyroid. 2009 Oct;19(10):1085-91. doi: 10.1089/thy.2009.0121. PMID 19803790
- [Background] Kovatcheva RD, Vlahov JD, Stoinov JI, Zaletel K. Benign Solid Thyroid Nodules: US-guided High-Intensity Focused Ultrasound Ablation-Initial Clinical Outcomes. Radiology. 2015 Aug;276(2):597-605. doi: 10.1148/radiol.15141492. Epub 2015 Mar 13. PMID 25768327
- [Background] Long B, Li L, Yao L, Chen S, Yi H, Ye X, Xu D, Wu P. Combined use of radioiodine therapy and radiofrequency ablation in treating postsurgical thyroid remnant of differentiated thyroid carcinoma. J Cancer Res Ther. 2015 Nov;11 Suppl:C244-7. doi: 10.4103/0973-1482.170530. PMID 26612446
- [Background] Palit TK, Miller CC 3rd, Miltenburg DM. The efficacy of thyroidectomy for Graves' disease: A meta-analysis. J Surg Res. 2000 May 15;90(2):161-5. doi: 10.1006/jsre.2000.5875. PMID 10792958
- [Background] Von Hofe SE, Dorfman SG, Carretta RF, Young RL. The increasing incidence of hypothyroidism within one year after radioiodine therapy for toxic diffuse goiter. J Nucl Med. 1978 Feb;19(2):180-4. PMID 627898
- [Background] Leslie WD, Ward L, Salamon EA, Ludwig S, Rowe RC, Cowden EA. A randomized comparison of radioiodine doses in Graves' hyperthyroidism. J Clin Endocrinol Metab. 2003 Mar;88(3):978-83. doi: 10.1210/jc.2002-020805. PMID 12629071
- [Background] Bartalena L, Baldeschi L, Dickinson A, Eckstein A, Kendall-Taylor P, Marcocci C, Mourits M, Perros P, Boboridis K, Boschi A, Curro N, Daumerie C, Kahaly GJ, Krassas GE, Lane CM, Lazarus JH, Marino M, Nardi M, Neoh C, Orgiazzi J, Pearce S, Pinchera A, Pitz S, Salvi M, Sivelli P, Stahl M, von Arx G, Wiersinga WM; European Group on Graves' Orbitopathy (EUGOGO). Consensus statement of the European Group on Graves' orbitopathy (EUGOGO) on management of GO. Eur J Endocrinol. 2008 Mar;158(3):273-85. doi: 10.1530/EJE-07-0666. No abstract available. PMID 18299459
- [Background] Wong KP, Lang BH, Ng SH, Cheung CY, Chan CT, Lo CY. A prospective, assessor-blind evaluation of surgeon-performed transcutaneous laryngeal ultrasonography in vocal cord examination before and after thyroidectomy. Surgery. 2013 Dec;154(6):1158-64; discussion 1164-5. doi: 10.1016/j.surg.2013.04.063. Epub 2013 Aug 19. PMID 23969288
- [Background] Philips Z, Bojke L, Sculpher M, Claxton K, Golder S. Good practice guidelines for decision-analytic modelling in health technology assessment: a review and consolidation of quality assessment. Pharmacoeconomics. 2006;24(4):355-71. doi: 10.2165/00019053-200624040-00006. PMID 16605282
- [Background] Metso S, Jaatinen P, Huhtala H, Luukkaala T, Oksala H, Salmi J. Long-term follow-up study of radioiodine treatment of hyperthyroidism. Clin Endocrinol (Oxf). 2004 Nov;61(5):641-8. doi: 10.1111/j.1365-2265.2004.02152.x. PMID 15521969
- [Background] Siebert U, Alagoz O, Bayoumi AM, Jahn B, Owens DK, Cohen DJ, Kuntz KM; ISPOR-SMDM Modeling Good Research Practices Task Force. State-transition modeling: a report of the ISPOR-SMDM Modeling Good Research Practices Task Force--3. Value Health. 2012 Sep-Oct;15(6):812-20. doi: 10.1016/j.jval.2012.06.014. PMID 22999130
- See also: Hong Kong Radiation Ordinance Chapter 303 — http://www.rbhk.org.hk/eng/ordin-cap303.html
- See also: Revisions to List of charges: G.N. 1488 to Gazette No. 12/2013 — http://www.gld.gov.hk/egazette/english/gazette/toc.php